CLINICAL TRIAL: NCT05298202
Title: The Influence of Topical Capsaicin on Thermoregulatory and Perceptual Outcomes During Exercise Within the Heat
Brief Title: The Influence of Capsaicin Gel During Exercise Within the Heat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0192-22-FB
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Acute Exercise; Heat Exposure
Keywords: heat exposure; exercise; capsaicin
MeSH Terms: conditions — Motor Activity | interventions — Capsaicin; Exercise

STUDY DESIGN:
Intervention Model Description: Each Subject acts as their own control in a repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Capsaicin gel application (Experimental): Capsaicin gel will be applied to the skin prior to exercise in the heat
  Interventions: Biological: Capsaicin; Other: Exercise; Other: Hot environment
- Hypoallergenic gel application (Placebo Comparator): A hypoallergenic gel will be applied to the skin prior to exercise in the heat
  Interventions: Biological: Control Gel; Other: Exercise; Other: Hot environment

INTERVENTIONS:
Biological: Capsaicin — application of capsaicin gel from shoulder to wrist and mid thigh to ankle
  Arms: Capsaicin gel application
Biological: Control Gel — application of hypoallergenic gel from shoulder to wrist and mid thigh to ankle
  Arms: Hypoallergenic gel application
Other: Exercise — treadmill walking 3.5 mph at 5% grade
Other: Hot environment — 38°C, 60% relative humidity

SUMMARY:
The purpose of this study is to examine the human thermoregulatory impact of applying a commercially available capsaicin gel to the skin prior to moderate intensity walking under heated conditions. Experimental Visits will consist of 30 min of treadmill walking at a moderate pace (3.5 mph, 5% grade) under hot conditions (38°C, 60%RH) and will be randomized and counterbalanced for capsaicin gel or a hypoallergenic gel (control) application.

Gels will be applied to areas commonly exposed during outdoor activity in warm conditions (shoulder to wrist, mid thigh to ankle). Accordingly, participants will wear shorts and a tank top shirt during exercise. Core temperature, skin temperature, galvanic skin response, laser doppler blood flow, and heart rate will be continuously recorded throughout the exercise bout via an integrated analog to digital converter. Sweat will be collected during exercise using commercially available absorbent patches. Thermal sensation will be assessed throughout exercise via the American Society of Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE) thermal sensation likert scale (cold to hot).

Lastly, nude body weight will be recorded pre and post exercise for sweat rate determination. The capsaicin and control trials will be separated by a 7-14 day washout period

DETAILED DESCRIPTION:
3 experimental visits to the laboratory will be conducted. All visits will take place at the University of Nebraska at Omaha, Exercise Physiology Laboratory. Visit 1 will consist of the physical activity readiness questionnaire (PARQ), adverse reaction to capsaicin, and body composition (hydrostatic weigh, bioelectrical impedance). Visits 2 and 3 will be separated by 7-14 days, randomized, and counterbalanced for experimental (capsaicin) and control (hypoallergenic cream) trials. Both the experimental and control visits will follow the same protocol.

Participants will arrive following an overnight fast state while also refraining from strenuous activity, alcohol consumption, tobacco use, and recreational drugs for the previous 24 hour period. During these visit researchers will apply capsaicin using a gloved hand from shoulder to wrist and mid thigh to ankle (areas outside of the clothing). A hypoallergenic cream will be applied during the control visit.

Exercise will consist of 30 min of moderate intensity treadmill walking (3.5 mph at 5% grade) within a heated temperature/humidity controlled chamber (38°C, 60% relative humidity). Participants will be weighed before, and after completion of the exercise calculate sweat rate. Prior to the exercise session, participants will sit for 5 min in an ambient room temperature environment as a baseline. During baseline and during the exercise core temperature, skin temperature, laser doppler blood flow, galvanic skin response, and heart rate will be collected continuously. Sweat patches will be adhered to the forehead during exercise at minute 10 for collection of sweat composition over the next 10-20 minutes. Thermal perception using the ASHRAE scale (cold to hot) will be assessed pre and during exercise.

EXPERIMENTAL VISIT 1 Visit 1 will take approximately 1 hour. Participants will then complete the physical activity readiness questionnaire (PARQ) to be cleared for physical activity. Participants will have a small amount of the capsaicin cream applied to a small area of the forearm (~2 x 2 in) to test for any adverse reaction over a period of 15 minutes. Those without a reaction will have height, weight, and body fat composition measured. Height and weight will be measured using a medical scale and stadiometer, respectively. Body fat will be assessed with hydrostatic weighing using an electronic load cell based system (Exertech, Dresbach, MN) correcting for residual lung volume or via a bio-electrical impedance analyzer (InBodyUSA, Cerritos, CA).

EXPERIMENTAL VISITS 2 AND 3 Visits 2 and 3 will take approximately 2 hours each. Upon arrival at the lab, a nude body weight will be collected with the subject in a private room. While still in the room, subjects will self-insert a rectal thermistor 12-15 cm beyond the anal sphincter and don a chest strap heart rate monitor. After dressing in their exercise clothing, subjects will exit the private room so that chest, forearm, and calf thermistors can be adhered to the skin with tape. Laser doppler flow (forearm and or/finger) will be adhered with tape and galvanic skin response (fingers) will be adhered using Velcro straps to the skin. Measuring instruments will be recorded using an integrated digital to analog converter (ADInstruments, Colorado Springs, CO).

Following instrumentation, subjects will sit for 5 minutes as a baseline in a temperate environment. Immediately after, a researcher with gloved hands will topically apply capsaicin or the control hypoallergenic cream from the shoulder to wrist and mid-thigh to ankle. Subjects will then enter the heat chamber (38°C, 60% relative humidity) and immediately begin a 30-minute walk on a treadmill (3.5 mph, 5% grade). Subjects will be intermittently asked to hold their arm steady for laser doppler flow collection (10, 20, 30 minutes). Subjects will also briefly pause at minute 10 in order to adhere an absorbent patch to their forehead for sweat collection over the following 10-20 minutes. Thermal perception using the ASHRAE scale (cold to hot) will be assessed pre and during exercise. After 30 minutes of walking, subjects will exit the chamber for removal of all skin and finger sensors. Subjects will then re-enter the private room, remove their own rectal thermistor with gloved hands, and then a final nude body weight will be recorded after toweling off.

The rectal thermistor will measure core temperature. The heart rate monitor will measure the beats of the heart. Skin thermistors will measure the temperature of the skin surfaces. Laser doppler flow measure the relative units of blood flow velocity. Galvanic skin response measures skin conductivity changes as individuals begin to sweat. Sweat is collected for assessment of sweat composition. Thermal perception is assessed for individual perception surrounding the temperature of the ambient environment. Nude body weight is measured to calculate sweat rate.

ELIGIBILITY:
Inclusion Criteria:

* 19-45 years of age
* cleared for physical activity via the 2022 physical activity readiness questionnaire (PARQ)
* no self-reported adverse reactions to capsaicin

Exclusion Criteria:

* outside 19-45 years of age
* not cleared for physical activity via the 2022 physical activity readiness questionnaire (PARQ)
* self-report or signs of sensitivity to capsaicin
* pregnant
* breast feeding

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin R Slivka, PHD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Capsaicin First (1 Day), Washout (7days) Then Hypoallergenic Gel (1 Day).: Capsaicin first, then hypoallergenic Gel.
  All participants will receive both Capsaicin and Control hypoallergenic cream (cross-over design ,randomized order, 7 days washout between) applied to the skin prior to exercise in the heat.
  both cremes were applied on the skin shoulder to wrist and mid-thigh to ankle.
- Hypoallergenic Gel First (1 Day), Washout (7 Days), Then Capsaicin (1 Day): hypoallergenic Gel first, then Capsaicin
  All participants will receive both Capsaicin and Control hypoallergenic cream (cross-over design ,randomized order, 7 days washout between) applied to the skin prior to exercise in the heat.
  both cremes were applied on the skin shoulder to wrist and mid-thigh to ankle.
Period: Overall Study
Arm/Group | Capsaicin First (1 Day), Washout (7days) Then Hypoallergenic Gel (1 Day). | Hypoallergenic Gel First (1 Day), Washout (7 Days), Then Capsaicin (1 Day)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants will receive both Capsaicin and Control hypoallergenic cream (randomized order, 7 days washout between) applied to the skin prior to exercise in the heat
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
Weight [Mean (Standard Deviation); unit: kg] | 86.2 (18.9)
Height [Mean (Standard Deviation); unit: cm] | 177.4 (6.7)
body fat [Mean (Standard Deviation); unit: percent body fat] | 20 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Skin Blood Flow
Description: Laser Doppler measurement of skin blood flow on the forearm. This is measured in arbitrary units where higher values represent higher blood flow.
Time Frame: 30 minutes into exercise bout
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
arbitrary units | 188.4 (104.9) | 139.2 (56.7)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority — time x treatment ANOVA; p = 0.284, ANOVA — difference between treatment and control

2. Primary Outcome: Sweat Composition
Description: Sodium concentrations in collected sweat
Time Frame: Final 10 minutes of the exercise bout (minutes 20-30 of exercise)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
mmol/L | 44.2 (16.4) | 47.5 (17.5)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority; p = .177, t-test, 2 sided

3. Primary Outcome: Sweat Rate
Description: To calculate sweat rate the difference in Nude body weight from pre to post exercise was measured (assuming weight loss is equal to sweat loss)
Time Frame: pre-post 30 minute exercise bout
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
Liters per hour | 1.23 (.37) | 1.43 (.43)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority; p = .122, t-test, 2 sided

4. Primary Outcome: Thermal Perception
Description: scale of thermal comfort developed by the American Society of Heating, Refrigerating and Air-Conditioning Engineers (ASHRAE). The ASHRAE is a 7-point scale to asses thermal sensation, which consists of seven verbal anchors: "cold (-3)", "cool (-2)", "slightly cool (-1)", "neutral (0)", "slightly warm (1)", "warm (2)", and "hot (3)". The score is reported as the value in "()"
Time Frame: at 30 minutes of exercise
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
score on a scale | 2.8 (.4) | 2.5 (.5)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority; p = .038, ANOVA; time x treatment anova

5. Primary Outcome: Average Skin Temperature
Description: average measurements from chest, forearm, and calf thermistors
Time Frame: at 30 minutes of the exercise bout
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
degrees C | 37.4 (.5) | 37.4 (.5)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority; p = .976, ANOVA

6. Primary Outcome: Core Temperature
Description: measured with rectal thermistor
Time Frame: at 30 minutes of the exercise bout
Measure: Mean (Standard Deviation); unit: degrees C
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
Number analyzed (Participants) | 12 | 12
degrees C | 37.8 (.6) | 37.8 (.5)
Statistical Analysis 1: Comparison: Capsaicin Gel Application vs Hypoallergenic Gel Application; Test type: Superiority; p = .747, ANOVA

ADVERSE EVENTS:
Time Frame: Through three visits, maximum of 29 days
Arm/Group | Capsaicin Gel Application | Hypoallergenic Gel Application
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05298202/Prot_SAP_000.pdf